CLINICAL TRIAL: NCT03871504
Title: Quantitative Sensory Testing, Physical Activity, and Body Composition in Adults
Brief Title: The Influence of Baseline Sensitivity and Expectation on Exercise-induced Hypoalgesia in Young Healthy Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marquette University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HR-2999
Record Dates: First submitted 2018-12-13; First posted 2019-03-12 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Healthy Subjects
Keywords: exercise; hypoalgesia; pain; expectation
MeSH Terms: conditions — Motor Activity; Pain

STUDY DESIGN:
Intervention Model Description: All subjects will participate in two randomized sessions (an exercise session and control session). The exercise session consists of submaximal isometric exercise while the quiet rest session consists of a rest for a period that mimics the time spent in exercise.
Who Masked: Participant
Masking Description: Participants are blinded to the hypothesis of this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- submaximal isometric exercise. (Experimental): submaximal isometric exercise will be performed.
  Interventions: Other: Submaximal isometric exercise
- Quiet rest. (No Intervention): Subject will rest in seating position for a period that mimics the exercise time.

INTERVENTIONS:
Other: Submaximal isometric exercise — The exercise is a submaximal isometric contraction
  Arms: submaximal isometric exercise.

SUMMARY:
The purpose of this study is to investigate the influence of baseline experimental pain sensitivity and expectation on the pain response following a single exercise session. Pain assessment will be done with different intensities of noxious stimuli. In addition, the expectation of how exercise impacts pain will be studied.

DETAILED DESCRIPTION:
The relation between baseline pain sensitivity and the pain response following exercise is not clear. The aims of this study are to investigate the influence of baseline experimental pain sensitivity on the pain response following submaximal isometric exercise, and whether expectations would influence outcomes with subsequent exposure to exercise.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* English proficiency

Exclusion Criteria:

* Acute pain condition
* Chronic pain condition
* Mental health disorder
* Cardiovascular disease
* Any chronic illness
* Difficulty with physical exercise
* Recent surgery
* Pulmonary disease
* Diabetes
* Smoking
* Raynaud disease
* Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2017-11-25 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
The change from baseline of pain ratings during temporal summation of pressure pain assessment | Before and immediately after exercise or quiet rest in session 1 and session 2 which will be on day 1 and day 7 of data collection.
  Temporal summation is the increase of pain over time caused by a constant or repetitive noxious stimulus. Pain reports will be obtained during the application of constant mechanical stimulus with various intensities. Subjects will be asked to rate the pain using a numerical pain rating scale that ranges from 0 (no pain) to 10 (worst pain). Pain ratings will be obtained at the beginning, during, and at the end of the test while a noxious stimulus is applied to the index finger. The change of pain ratings relative to baseline after exercise or quiet rest will be assessed.

SECONDARY OUTCOMES:
Expectation | Before exercise which will be on day 1 and day 7 of data collection.
  Subjects will be asked about their expectation of whether exercise will increase, decrease, or have no effect on the pain.
State version of the State-Trait Anxiety Inventory (STAI) | After each temporal summation protocol in the first and second session which are on day 1 and day 7 of data collection.
  A 20-item questionnaire from state-trait anxiety inventory that evaluates different feelings the subject may or may not have at the moment. The score of the questionnaire ranges from 0 to 80. Higher scores indicate greater state anxiety levels.
Trait version of the State-Trait Anxiety Inventory (STAI) | Baseline (beginning of session 1) which is day 1 of the data collection.
  A 20-item questionnaire from state-trait anxiety inventory that evaluates how the subject feels in general and not restricted to the current moment. The score of the questionnaire ranges from 0 to 80. Higher scores indicate greater trait anxiety levels.
Pain catastrophizing scale | Baseline (beginning of session 1) which is day 1 of the data collection.
  A 13-item scale that evaluates if the subject has an exaggerated negative mental set towards pain. It has 3 sub-scales which are magnification, rumination, and helplessness. The scores of the sub-scales are summed to get the total score. The total score ranges from 0 to 52. Greater scores indicate greater catastrophizing thinking.
Situational pain catastrophizing scale | After each temporal summation protocol in the first and second session which are day 1 and day 7 of data collection.
  A 6-item questionnaire that explores the negative mental set or catastrophizing thinking in reference to a particular experimental pain experience (i.e., temporal summation protocol). The score ranges from 0 to 24 with higher scores indicating greater situational catastrophizing.
Physical activity assessment using International physical activity questionnaire. | Baseline (beginning of session 1 or 2) which is either day 1 or day 7 of data collection.
  International physical activity questionnaire (IPAQ) will be used to assess physical activity in the past week. IPAQ evaluates physical activity not only related to leisure time but also related to other domains such as transportation, work, gardening or house related physical activities. The questionnaire has been shown to be reliable and valid. The time spent in moderate to vigorous physical activity (minutes/ week) from every domain will be summed with 0 indicating no time (minutes / week) spent moderate to vigorous activities and higher values indicate greater time spent in moderate to vigorous physical activity.
Muscle mass assessment using Dual-energy x-ray absorptiometry. | Baseline (in the first or second session) which is either day 1 or day 7 of data collection.
  Dual-energy x-ray absorptiometry (General Electric Healthcare, Madison, Wisconsin) is an x-ray scan that is used to assess muscle mass.
Fat mass assessment using Dual-energy x-ray absorptiometry. | Baseline (in the first or second session) which is either day 1 or day 7 of data collection.
  Dual-energy x-ray absorptiometry (General Electric Healthcare, Madison, Wisconsin) is an x-ray scan that is used to assess fat mass.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Hoeger Bement, PT, PhD, Principal Investigator — Marquette University
Locations (1):
- Marquette University, Milwaukee, Wisconsin, United States